CLINICAL TRIAL: NCT03167567
Title: The Effect of Medical Clowning on Primipara Women During Labor
Brief Title: The Effect of Medical Clowning During Labor
Acronym: MedClown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Izhar Ben Shlomo, Professor, The Baruch Padeh Medical Center, Poriya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0081-15-POR
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Mental Status Change; Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Women who will agree to be escorted by a medical clown during their first labor will be interviewed after delivery regarding their experience. Their answers will be compared to those of women whe were not escorted by a clown.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): These women will have a medical clown present in the room during their labor
  Interventions: Behavioral: Presence of a medical clown during labor
- Control (No Intervention): These women will not have a medical clown in the room during their labor

INTERVENTIONS:
Behavioral: Presence of a medical clown during labor — Presence of a medical clown during labor
  Arms: intervention

SUMMARY:
Women during their first labor will be offered the assistance of a medical clown. Their experience will be compared after delivery with that of primiparae who were not helped by a medical clown.

DETAILED DESCRIPTION:
Introduction Midwives have been known for many years to give support, care and advice to pregnant women during pregnancy, birth and after birth. The word midwife literally means 'with woman'. It is known that throughout the age's women during childbirth depended upon a skilled person (usually a woman in the olden days). Her skill is based partly on art and partly on science. Art: the ability to understand the woman's need, encourage and build her confidence. Science: knowledge and decision-making. The midwife refrains from taking control away from the mother, but is at hand to step in where assistance is needed (Myles 1999).

Literature review Labor is a normal physiological process, but is usually associated with pain and discomfort. (Othman, Jones, & Neilson, 2012). Over the years, various measures to relieve stress, discomfort, pain, fear and anxiety during labor have been explored. (Ganji, shirvani, rezaei-Abhari, & Danesh, 2013). Therefore, these issues that impact the wellbeing of the pregnant and laboring woman are of primary interest and value to caregivers. (Bergstrom, Kieler, & Waldenstrom, 2009). However, many women would like to have a choice in pain relief during labor and also would like to avoid invasive methods of pain management in labor. (Klomp, van Poppel, Jones, Lazet, Di Nisio, & Lagro-Janssen, 2012). Adams, Eberhard-Gran, and Eskild, (2012) concluded that duration of labor was longer in women with fear of childbirth than in women without it. The search for supporting measures such as the use of birthing in water, yoga, and other non invasive approaches in addition to drug administration during labor is crucial.

Midwives support natural birth as much as possible. Thus, preparation classes have been introduced to teach and enlighten pregnant woman, in order for them to understand the changes and process of pregnancy, labor and after birth concerning their bodies. Stress, depression, and anxiety affect 15 to 25% of pregnant women. However, fewer than 20% of prenatal care providers assess and treat mental health problems and fewer than 20% of pregnant women seek mental healthcare (Kingston. D. et al., 2014).

In The Baruch Pade Medical Center there are approximately 60 live births of primiparous women monthly.

Medical clowning has been used as a supportive factor, mostly in pediatric settings (Gorfinkle et al., 1998; Koller & Gryski, 2008; Scheyer et al., 2008). Medical clowns are trained professionals (Bornstein, 2008; Hart, 2012) who master at least one of the various stage arts such as theatre, acting, circus or puppetry. Their aim is to improve the mental and physical well-being of patients by easing pain and anxiety due to hospitalization. The clowns strive to be an integral part of the medical team and are even present during physically intrusive procedures (Hart, 2012; Smerling et al., 1999; Tener, Lnag-Franco, Ofir & Lev-Wiesel, 2012). The medical clown plays a therapeutic and a diagnostic role and is perceived as any other paramedical therapist (Hart, 2012).

The medical clown uses a broad spectrum of verbal and non-verbal artistic tools including mime, movement, play, act and music in order to create humor and an alternative, imaginative safe reality (Nuttman-Schwartz, Scheyer & Tzioni, 2010). By doing so, the clown builds an empowering and supportive relationship (Bornstein, 2008; Koller & Gryski, 2008 The empirical data regarding medical clowns in hospitals is limited (e.g. Battrick, Glasper & Weaver, 2007; Bornstein, 2008; Weaver, Prudhome, Battrick & Glasper, 2007). However, the influence of humor and laughter on decreasing anxiety levels while preparing for surgery, post fertility treatments, children undergoing intra-articular corticosteroid injection, children with special needs and sexually abused children has been studied (Fernandes & Arriaga, 2010; Friedler et al., 2010; Higueras et al., 2006; Kingsnorth, Blain & McKeever, 2010; Koller & Gryski, 2008; Tener et al., 2010, 2012; Oren-Ziv, Hanuka, Rotchild, Gluzman, & Uziel, 2012; Vagnoli, Caprilli & Messeri, 2010; Vagnoli, Caprilli, Robiglio & Messeri, 2005). Additional studies found that medical clowns are helpful both for health care providers (Smerling et al., 1999) and patients (Battrick et al., 2007) with no difference between hospitalized patients and outpatients (Scheyer et al., 2008; Weaver et al., 2007).

Medical clowns have been introduced into the hospital settings in the pediatric settings, IVF, operating theaters, oncology, geriatrics and others with positive results shown statistically. The benefits of medical clowning intervention, are in encouraging and supporting patients to co-operate with treatment procedure, in reducing stress, coping with fears, anxiety and reducing pain.

Extensive evidence indicates that negative and positive affective traits such as depression, worry, calmness, or cheerfulness can influence physical health (Papousek & Schulter, 2008). Also, There is strong evidence that positive and negative affects strongly influence subjective physical health (such as symptom reporting, self rated health or perception of the examinations performed) (Cohen, Doyle, Turner, Alper & Skoner, 2003; Cohen 1995; Hirdes & Forbes, 1993; Watson & Pennebaker, 1989). An increase in the patient wellbeing could be the result of an increase in positive affect, a decrease in negative affect, or a combination of the two factors (Charles, Reynolds & Gatz, 2001). A number of methods are used to induce positive moods and reduce negative affect in the experimental studies of mood and health. In Pressman and Cohen (2005, 2006) review of 45 empirical studies about affect and health, manipulations that involved active participation or were particularly engaging to the participant were found to be more effective in influencing positive and negative affect, whereas more passive manipulations failed to do so. Medical Clowns may be an active and engaging way of enhancing the positive and reducing the negative affect regarding primiparas.

In the delivery room there are women in different stages of labor that are anxious and fearful. It is to be noted that medical clowns have been working at The Padeh Medical Center for the past 10 years and the area is still expanding to different departments in the hospital such as: high risk pregnancy, parents in the neonatal intensive care units (NICU) and in the In Vitro fertilization (IVF) unit. In addition, following a meeting of women undergoing IVF treatments and women hospitalized due to high risk pregnancies, we have been contacted by several women who expressed their wish to have a medical clown present during their delivery. With this enlightenment, we find it necessary to check if it is possible to assist the birthing woman and her care givers in the labor room with medical clowning in the birth process.

The purposes of this study are:

1. To study the effect of female medical clowns on relieving anxiety during labor
2. To document whether the use of medical clowning can reduce the time for use of pain relievers and shorten the duration of labor.

Methods:

Before their first birth, while visiting the hospital, a questionnaire will be administered to the women. This will be a Likert-type response scale ranging from 1 (Not at all) to 5 (the most) rated by the primiparas, examining the women's perception of incorporating medical clowning in the labor process. After birth, PANAS Scales short questionnaires which measure the positive and negative affect of the primiparas will be filled in by the women within 48 hours after giving birth (Charles, Reynolds & Gatz, 2001; Watson & Clark, 1988). In addition, we will record measures regarding the length of labor and at what stage/after after entering the labor room women asked for analgesics, what kind of analgesics they asked for, and when and what did they receive.

Patients:

Two hundred women, older than 18 years, at their first expected labor,100 as intervention group and 100 as the control group.

1. A candidate who will arrive at The Padeh Medical Center will be approached by a midwife or a doctor with information about the research and will be asked if she wishes to take part.
2. According to the patients' request and to the clown's shift, the patients will be recruited to either the control or the research group.
3. A research team member will inform the participants who will be allocated to the intervention that they can, at any stage, ask the clown to leave the delivery room. In addition, primiparas from both groups will be informed that they can at any stage ask to be excluded from the research. All these will be also explicitly stated in the consent form which she will sign. Each participant will receive a number and her details will be kept and available to the staff members only.
4. The delivery room staff will guide the clown as to when to join the primipara in the delivery room. The medical clown will enter the delivery room and stay with the woman as long as she wishes (within the clown's shift of 3 hours).
5. After the delivery a member of the research team or a research assistant will fill in the demographic questionnaire.
6. Within 48 hours after delivery the patient will fill in the PANAS questionnaire.
7. At the conclusion of all the above, all data regarding the delivery, drug usage and length of labor, complications if any will be entered to the CRF with all other patients' data.

Clowns:

The female medical clowns will be present in the delivery rooms for a shift of 3 hours twice a week.

Research tools:

1. Likert-type scale questionnaire (appendix 1).
2. Demographic questionnaire for the primiparas. (Appendix 2)
3. The PANAS scale - brief measures of positive and negative affect (appendix 3). Will be given to the research group.
4. The PANAS scale - brief measures of positive and negative affect (appendix 3). Will be given to the control group.
5. Information from the reports of the labor department regarding the length of labor and of the analgesics requested by (timing and kind) given to the women and any complications will be documented.

Data analysis:

Data from the Likert-type scales questionnaire will be analyzed in order to capture the perception of women before labor of introducing medical clowns during labor. Data from the PANAS questionnaire will be analyzed. Negative and Positive affect will be assessed in adapted scales. Separate Hierarchical Multiple Regression analyses will be conducted to examine the influence of the medical clown in the two dependent variables: Positive and Negative affect. In addition, we will try to understand what parameters from the demographic questionnaire effect the primipara's reaction and co-operation with the medical clown during labor.

Control of Potential Biases:

The research group will contain two medical clowns, a gynecologist and 2 RN midwifes from the labor ward team who have almost no experience in working with medical clowns and has no preconception about the issue.

References Adams, S., Eberhard-Gran, M. and Eskild, A. (2012), Fear of childbirth and duration of labour: a study of 2206 women with intended vaginal delivery. BJOG: An International Journal of Obstetrics & Gyneacology, 119: 1238-1246 Battrick, C., Glasper, E. A., Prudhoe, G., & Weaver, K. (2007). Clown humour: The perception of doctors, nurses, parents and children. Journal of Children's and Young People's Nursing, 1(4), 174-179.

Bennett, V. R., and Brown, L. K. (1999), Myles Textbook for Midwives, 13th edn. Churchill Livingstone.

Bergstrom, M., Kieler, H. and Waldenstom, U. (2009), Effects of natural childbirth preparation versus standard antenatal education on epidural rates, experience of childbirth and parental stress in mothers and fathers: a randomized controlled multi center trial. BJOG: An International Journal of Obstetrics & Gynecology, 116:1167-1176. doi: 10.1111/j.1471-0528.2009.02144.x Bornstein, Y. (2008). Medical clowns at hospitals and their effect on hospitalized children. Harefuah, 147(1), 30-32.

Carstensen, L. L., Pasupathi, M., Mayr, U., & Nesselroade, J. (2000). Emotion experience in everyday life across the adult life span. Journal of Personality and Social Psychology, 79, 644-655.

Charles, S.T., Reynolds, C.A., & Gatz, M. (2001). Age-related differences and change in positive and negative affect over 23 years. Journal of personality and social psychology 80(1), 136-151. doi:10.1037/0022-3514.80.1.136 Cohen, S., Doyle, J.W., Turner, R. B., Alper, C.M. & Skoner, D. (2003). Emotional style and susceptibility to the common cold. Journal of Psychosomatic Medicine. 65(4), 652-657.

Cohen, S., & Pressman, S. D. (2006). Positive affect and health. Current Directions in Psychological Science, 15(3), 122-125.

Denzin, N.K., & Lincoln, Y.S. (1994). Handbook of qualitative research. Thousand Oaks, CA: Sage.

Fernandes, S. C., & Arriaga, P. (2010). The effects of clown intervention on worries and emotional responses in children undergoing surgery. Journal of Health Psychology, 15, 405-415. doi:10.1177/1359105309350231 12 Friedler, S., Glasser, S., Azani, L., Freedman, L. S., Raziel, A., Strassburger, D., Ron-El, R., & Lerner-Geva, L. (2011). The effect of medical clowning on pregnancy rates after in vitro fertilization and embryo transfer (IVF-ET). Fertility and Sterility, 95(6), 2127-2130. doi:10.1016/j.fertnstert.2010.12.016 Ganji, Z., Shirvani, M. A., Rezaei-Abhari, F. and Danesh, M. (2013), The effect of intermittent local heat and cold on labor pain and child birth outcome. Iranian Journal of Nursing and Midwifery Research. Jul-Aug; 18(4): 298-303.

Gorfinkle, K. S., Slater, J. A., Bagiella, E., Tager, F. A., & Labinsky, E. B. (1998). Child behavioral distress during invasive oncologic procedures and cardiac catheterization with the big apple circus clown care unit. Pediatric Research, 43(4), 12. doi:10.1203/00006450-199804001-00076 Hanuka, P., Rotchild, M., Gluzman, A. and Uziel, Y. (2011), Medical clowns: dream doctors as an important team member in the treatment of young children with juvenile idiopathic arthritis. Pediatric Rheumatology, 9(suppl 1):p118 Hart, J. (2012). Not just clowning around: Medical clowns in health care teams: An interview with Arthur I. Eidelman, MD. Alternative and Complementary Therapies, 18(6), 319-323. doi:10.1089/act.2012.18602 Higueras, A., Carretero-dios, H., Munoz, J. P., Idni, E., Ortiz, A., Rinkon, F., & Prieto- Merino, D. (2006). Effects of humor-centered activity on disruptive behavior in patients in a general hospital psychiatry ward. International Journal of Clinical and Health Psychology, 6, 53-64.

Hirdes, J.P. & Forbes, W.F. (1993). Factors associated with the maintenance of good self-rated health. Journal of Aging and Health. 5(1), 101-122.

Kingsnorth, S., Blain, S., & McKeever, P. (2010). Physiological and emotional responses of disabled children to therapeutic clowns: A pilot study. Retrieved from February 4, 2010, from http://creativecommons.org/licenses/by-nc/2.5. doi.org/10.1093/ecam/neq008 Kingston, D., Austin, MP., Hegadoren, K., McDonald, S., Lasiuk, G., McDonald, S., Heaman, M,. Biringer, A., Sword, W., Giallo, R., Patel, T., Lane-Smith, M., van Zanten, SV. (2014), Study protocol for a randomized, controlled, superiority trial comparing the clinical and cost- effectiveness of integrated online mental health assessment-referral-care in pregnancy to usual prenatal care on prenatal and postnatal mental health and infant health and 13 development: the Integrated Maternal Psychosocial Assessment to Care Trial (IMPACT). Trials. Mar 6;15(1):72.[Epub ahead of print] Klomp, T,. van Poppel M., Jones L,. Lazet J., Di Nisio, M., Lagro-Janssen, AL. (2012), Inhaled analgesia for pain management in labour. Cochrane Database Syst Rev. Sep 12(9):CD009351.doi: 10.1002/14651858.CD009351.pub2.

ELIGIBILITY:
Inclusion Criteria:

* All planned vaginal first delivery
* Older than 18 years
* Younger than 40 years
* Mentally healthy

Exclusion Criteria:

* Previous known mental disorder
* Younger than 18 years
* Older than 40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Mood and recollection of experience | Women will be interviewed within the immediate 48 hours post partum
  Structered interview

CONTACTS AND LOCATIONS:
Overall Officials: Odelia Katz, PhD, Study Chair — CEO Research Authority

IPD SHARING:
Plan to Share IPD: No